CLINICAL TRIAL: NCT02215278
Title: A Multiple Meal Stable Iron Isotope Study in Iron Deficient Rwandese Women to Investigate the Performance of Low Phytic Acid Bean Seeds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GroundWork (Other)
Collaborators: HarvestPlus (Other)
Responsible Party: Principal Investigator, Nicolai Petry, Dr. of Science ETH, GroundWork
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: lpa_002
Record Dates: First submitted 2014-06-12; First posted 2014-08-13 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Enrichment of Blood With Stable Iron Isotopes
Keywords: iron biofortification; lpa bean; stable iron isotope study; phytic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- low phytic acid bean (lpa variety) (Experimental)
  Interventions: Dietary Supplement: 10 x 55 g/ bean per arm
- high iron biofortified bean variety (Experimental)
  Interventions: Dietary Supplement: 10 x 55 g/ bean per arm
- normal iron, normal phytic acid bean (Experimental)
  Interventions: Dietary Supplement: 10 x 55 g/ bean per arm

INTERVENTIONS:
Dietary Supplement: 10 x 55 g/ bean per arm

SUMMARY:
Recent iron absorption studies with biofortified beans indicated that the currently developed beans do not provide an extra amount of iron compared to normal iron beans. This effect was ascribed to the inhibitory nature of phytic acid (PA), which is present in high concentrations. A possible solution to alleviate problems associated with the high PA concentration in beans might be low phytic acid (lpa) bean seeds. These beans, which exhibit a good agronomic performance, were tested in a human absorption study in Switzerland and provided a higher amount of bioavailable iron compared to their parent beans with normal PA concentrations. However, the informative value of the study for the real life situation is limited due to the simple study design with a relatively large amount of isotopic label added extrinsically (≈30% of total iron). Furthermore, the study was conducted in iron sufficient women in a non-bean consuming population. Additional investigations are necessary to verify that iron bioavailability from lpa beans is high and that their performance is better compared to common biofortified beans in a real life situation. A multiple meal randomized crossover study in Rwandese women with low iron status will be done to measure iron absorption from three different beans (lpa bean line, biofortified high iron bean, normal iron bean as a control). During the study, the subjects will receive multiple meals to reduce the amount of extrinsic label, therefore more closely simulating hypothetical dietary iron intake from lpa beans. This will also allow to avoid an overestimation of the effect of inhibitors and to minimize the influence of intra subject day to day variation. The study will be divided into two parts. In part one, two of the three bean varieties will be fed as part of composite meals over several days (morning and lunch) and in part two, the remaining bean will be administered as part of composite meals over several days (morning and lunch). Iron absorption from the three varieties will be measured and compared with erythrocyte incorporation of stable isotopic labels 14 days after test meal administration.

ELIGIBILITY:
Inclusion Criteria:

* non pregnant women, non lactating women
* 18-30 years
* <65 kg

Exclusion Criteria:

* metabolic, chronic or gastrointestinal disease
* long term medication
* blood donation within the last 6 month

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Iron bioavailability from lpa bean variety compared to an iron biofortified variety | 2 month
  Iron bioavailability is determined by measuring the amounts of isotopic labels in blood 14 d after administration of the test meals. It is calculated on the basis of the shift in iron isotope ratios and on the estimated amount of iron circulating in the body. Circulating iron is calculated based on the blood volume estimated from height and weight and measured Hb concentration. The calculations are based on the principles of isotope dilution. For calculation of fractional absorption, 80% incorporation of the absorbed Fe into red blood cells is assumed.
  Isotopic analysis are performed by negative thermal ionization mass spectrometry using a magnetic sector field mass spectrometer equipped with a multi-collector system for simultaneous ion beam detection

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Petry, PhD, Principal Investigator — GroundWork; Diego Moretti, PhD, Principal Investigator — ETH Zurich
Locations (1):
- University of Rwanda, Butare, Huye, Rwanda

REFERENCES:
- [Derived] Petry N, Rohner F, Gahutu JB, Campion B, Boy E, Tugirimana PL, Zimmerman MB, Zwahlen C, Wirth JP, Moretti D. In Rwandese Women with Low Iron Status, Iron Absorption from Low-Phytic Acid Beans and Biofortified Beans Is Comparable, but Low-Phytic Acid Beans Cause Adverse Gastrointestinal Symptoms. J Nutr. 2016 May;146(5):970-5. doi: 10.3945/jn.115.223693. Epub 2016 Mar 30. PMID 27029940